CLINICAL TRIAL: NCT03465904
Title: A Phase III Randomized, Double-blind, Sham-controlled Trial of e-TNS for the Acute Treatment of Migraine (The TEAM Study)
Brief Title: A Phase III Trial of e-TNS for the Acute Treatment of Migraine
Acronym: TEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cefaly Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 51401
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Results first posted 2019-07-01 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Verum (Experimental): 2-hour external trigeminal nerve stimulation with the Verum Cefaly® Abortive Program device, as abortive treatment of an early stage migraine attack
  Interventions: Device: Verum Cefaly® Abortive Program device
- Sham (Sham Comparator): 2-hour external trigeminal nerve stimulation with the Sham Cefaly® Abortive Program device, as abortive treatment of an early stage migraine attack
  Interventions: Device: Sham Cefaly® Abortive Program device

INTERVENTIONS:
Device: Verum Cefaly® Abortive Program device — The Cefaly® Abortive Program device is an external cranial neurostimulator designed for supraorbital neurostimulation, also known as external Trigeminal Nerve Stimulation (e-TNS). The Verum Cefaly® Abortive Program device will deliver verum external trigeminal nerve stimulation.
  Arms: Verum
Device: Sham Cefaly® Abortive Program device — The Cefaly® Abortive Program device is an external cranial neurostimulator designed for supraorbital neurostimulation, also known as external Trigeminal Nerve Stimulation (e-TNS). The Sham Cefaly® Abortive Program device will deliver sham external trigeminal nerve stimulation.
  Arms: Sham

SUMMARY:
The main objective of this study is to have Phase III evidences of the efficacy of the Cefaly® Abortive Program device used at home for 2 hours to treat a migraine attack. This randomized, double-blind, sham-controlled trial will study the abortive treatment of migraine using the Cefaly® Abortive Program device.

DETAILED DESCRIPTION:
The main objective of this study is to have Phase III evidences of the efficacy of the Cefaly® Abortive Program device used at home for 2 hours to treat a migraine attack, as triptans are generally used. That is to say having randomized, double-blind, sham-controlled data of the efficacy and safety of the Cefaly® Abortive Program device in the abortive treatment of acute migraine as measured by 2-hour pain freedom, pain relief and migraine-associated symptoms freedom, plus evolution of these measurements for 24 hours after the beginning of the treatment session.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 65 on the day of signing the informed consent form
2. ≥ 1-year history of migraine with or without aura according to the diagnostic criteria listed in International Classification of Headache Disorders (ICHD)-3 beta (2013) section 1, migraine, with the exception of aura without headache, hemiplegic migraine and brainstem aura migraine
3. Migraine onset before the age of 50
4. Having between 2 and 8 moderate or severe migraine attacks (Grade 2 or 3) per month in each of the two months prior to screening
5. Patient understands the study procedures, alternative treatments available, and voluntarily agrees to participate in the study by giving written informed consent
6. Patient is able to read and understand the written information (instruction sheet, paper diary and Adverse Events reporting form)

Exclusion Criteria:

1. Patient has difficulty distinguishing his/her migraine attacks from tension-type headaches
2. Patient has more than 15 headache days per month
3. Patient having received supraorbital nerve blocks in the prior 4 months
4. Patient having received Botox treatment in the prior 4 months
5. Modification of a migraine prophylaxis treatment in the previous 3 months
6. Diagnosis of other primary headache disorders, except rare (< 4) tension-type headaches per month
7. Diagnosis of secondary headache disorders including Medication Overuse Headache (MOH)
8. Patient abusing opioids or user of recreational or illicit drugs or having had a recent history (within the last year) of drug or alcohol abuse or dependence
9. Implanted metallic or electronic device in the head
10. Cardiac pacemaker or implanted or wearable defibrillator
11. Patient having had a previous experience with the Cefaly® device
12. Migraine Aura without headache
13. Patient is currently participating or has participated in a study with an investigational compound or device in the last 30 days before the screening visit (Visit 1)
14. Patient not having the ability to use appropriately the device and/or to perform himself/herself or bear the first 20-minute stimulation session during the training test session at the study site

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deena Kuruvilla, M.D., Principal Investigator — Yale University
Locations (10):
- United States (10):
  - Clinical Research Consortium, Tempe, Arizona
  - Pharmacology Research Institute, Encino, California
  - Yale University, New Haven, Connecticut
  - Palm Beach Research Center, West Palm Beach, Florida
  - Meridian Clinical Research (Savannah Neurology), Savannah, Georgia
  - Meridian Clinical Research (Rockville Neurology), Rockville, Maryland
  - Clinical Research Consortium, Las Vegas, Nevada
  - Rochester Clinical Research, Rochester, New York
  - Rapid Medical Research Inc., Cleveland, Ohio
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuruvilla DE, Mann JI, Tepper SJ, Starling AJ, Panza G, Johnson MAL. Phase 3 randomized, double-blind, sham-controlled Trial of e-TNS for the Acute treatment of Migraine (TEAM). Sci Rep. 2022 Mar 24;12(1):5110. doi: 10.1038/s41598-022-09071-6. PMID 35332216

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 10, 2018 and January 11, 2019, 626 subjects were screened for eligibility, and 607 were enrolled across ten centers in the United States.
Period: Overall Study
Arm/Group | Verum | Sham
Started | 299 | 308
Completed | 259 | 279
Not Completed | 40 | 29
Not completed — Withdrawal by Subject | 9 | 5
Not completed — Lost to Follow-up | 11 | 9
Not completed — Protocol Violation | 20 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Verum | Sham | Total
Number analyzed (Participants) | 259 | 279 | 538
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.22 (11.62) | 42.0 (12.30) | 41.14 (12.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214 | 229 | 443
  Male | 45 | 50 | 95
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Migraine type [Count of Participants; unit: Participants]
  Migraine with aura | 113 | 111 | 224
  Migraine without aura | 146 | 168 | 314
Headache pain severity [Count of Participants; unit: Participants]
  No Pain | 1 | 0 | 1
  Mild Pain | 1 | 0 | 1
  Moderate pain severity | 155 | 166 | 321
  Severe pain severity | 102 | 113 | 215
Most Bothersome Symptom [Count of Participants; unit: Participants]
  Nausea as MBS | 55 | 54 | 109
  Vomiting as MBS | 4 | 7 | 11
  Sensitivity to light as MBS | 162 | 183 | 345
  Sensitivity to sound as MBS | 38 | 35 | 73
Migraine Associated Symptom [Number; unit: occurrences reported by subjects]
  Photophobia | 247 | 259 | 506
  Phonophobia | 207 | 228 | 435
  Nausea | 169 | 172 | 341
  Vomiting | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Pain Freedom at 2 Hours
Description: The percentage of patients having a reduction of a moderate or severe migraine headache (Grade 2 or 3) at baseline to no headache (Grade 0) at 2 hours after the beginning of the e-TNS session.
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Verum | Sham
Number analyzed (Participants) | 259 | 279
Participants | 66 | 51

2. Primary Outcome: Most Bothersome Migraine-associated Symptom Freedom at 2 Hours
Description: The percentage of patients with absence, at 2 hours after the beginning of the e-TNS session, of the most bothersome migraine-associated symptom identified at baseline.
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Verum | Sham
Number analyzed (Participants) | 259 | 279
Participants | 146 | 118

3. Secondary Outcome: Pain Relief at 2 Hours
Description: The percentage of patients having a reduction of a moderate or severe migraine headache (Grade 2 or 3) at baseline to a mild headache or to no headache (Grade 1 or 0) at 2 hours after the beginning of the e-TNS session.
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Verum | Sham
Number analyzed (Participants) | 259 | 279
Participants | 180 | 154

4. Secondary Outcome: Percentage of Patients With Absence of Photophobia, Phonophobia, Nausea, Vomiting at 2 Hours
Description: The percentage of patients with absence of photophobia, phonophobia, nausea, vomiting at 2 hours after the beginning of the e-TNS session.
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Verum | Sham
Number analyzed (Participants) | 259 | 279
Participants | 110 | 95

5. Secondary Outcome: Use of Rescue Medication Between 2 and 24 Hours
Description: The percentage of patients who took anti-migraine rescue medication between 2 and 24 hours after the beginning of the e-TNS session.
Time Frame: 2-24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Verum | Sham
Number analyzed (Participants) | 209 | 237
Participants | 82 | 105

6. Secondary Outcome: Sustained Pain Freedom at 24 Hours
Description: The percentage of patients having no headache (Grade 0) at 2 hours, with no use of anti-migraine rescue medication and no relapse of headache pain within the 24 hours after the beginning of the e-TNS session.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Verum | Sham
Number analyzed (Participants) | 259 | 279
Participants | 59 | 44

7. Secondary Outcome: Sustained Pain Relief at 24 Hours
Description: The percentage of patients having mild or no headache (Grade 1 or 0) at 2 hours, with no use of anti-migraine rescue medication and no relapse of headache pain within the 24 hours after the beginning of the e-TNS session.
Time Frame: 2-24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Verum | Sham
Number analyzed (Participants) | 259 | 279
Participants | 119 | 96
Statistical Analysis 1: Comparison: Verum vs Sham; Identical statistical analyses were performed for the intent-to-treat (ITT) and the per protocol (PP) populations. The ITT population consisted of all randomized patients, who received any duration of sham or verum treatment and returned completed study materials. The PP population consisted of patients who strictly met inclusion criteria and completed at least 60 min of treatment; Test type: Superiority — Our power analysis indicated that a minimum of 239 patients per group was needed to provide 90% power to detect a 13.4% difference in the primary outcome, pain freedom at 2 h. Accounting for an estimated attrition rate of 20%, we aimed to enroll 299 patients per group; p < 0.05, Chi-squared — All analyses were performed using SPSS, version 26.0 with two-sided levels of statistical significance established at p < 0.05; A Chi-square test of independent proportions was used to compare primary and secondary efficacy outcomes between groups

ADVERSE EVENTS:
Time Frame: The data was collected during the 24 hours following the beginning of the treatment
Arm/Group | Verum | Sham
All-Cause Mortality (participants affected / at risk) | 0/298 | 0/303
Serious Adverse Events (participants affected / at risk) | 0/298 | 1/303
Other Adverse Events (participants affected / at risk) | 22/259 | 8/279
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Verum (N=298) | Sham (N=303)
Appendicitis leading to appendectomy (Surgical and medical procedures) | 0 (0) | 1 (1) — This Serious Adverse Event was not related to the subject's participation in the study and was not reportable neither to the Institutional Review Board (IRB) nor to the FDA (the subject did not apply the treatment).
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Verum (N=259) | Sham (N=279)
Forehead paresthesias, discomfort, or burning (Nervous system disorders) | 9 (9) | 1 (1) — Expected side effect of the Cefaly® device
Nausea / Vomiting (Nervous system disorders) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Neck Stiffness / Muscle tension (Nervous system disorders) | 1 (1) | 2 (2)
Worsened Headache (Nervous system disorders) | 2 (2) | 0 (0)
Orodynia - tooth or jaw pain (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Restlessness (Nervous system disorders) | 1 (1) | 1 (1)
Abdominal Discomfort or Cramping (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Dry Mouth (Nervous system disorders) | 1 (1) | 0 (0)
Excessive Sweating (Nervous system disorders) | 2 (2) | 0 (0)
Sleepiness / Sedation (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of 90 days from the time submitted to the sponsor for review. Sponsor may request:

* deletion of any trade secret, proprietary, or confidential information of Sponsor
* an additional 90 days to take measures to preserve its Intellectual Property rights

Sponsor's written consent is required for results communication before trial completion.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/04/NCT03465904/Prot_SAP_000.pdf